CLINICAL TRIAL: NCT01641874
Title: The McKenzie System's Derangement Classification in Osteoarthritic Knees: Efficacy of McKenzie Treatment Versus Evidence Based Care: A Randomised Controlled Trial
Brief Title: The McKenzie System With Arthritic Knees: Do Some Knees Respond to Specific Exercise More Than General or no Exercise
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Richard Rosedale, Physiotherapist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16399E; IMDTRF (Other Grant/Funding Number: IMDTRF)
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; McKenzie system; Exercise; Mechanical Diagnosis and Therapy; Directional preference
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Specific directional exercise (Experimental): During the assessment a specific exercise will be identified for this group. The exercise will consist of a repeated specific end range movement of the knee
  Interventions: Procedure: Exercise
- Evidence based exercise (Active Comparator): Quadriceps strengthening and advice on aerobic exercises will be given
  Interventions: Procedure: Evidence based exercise
- No intervention (No Intervention): Patient waits on the surgeons waiting list for next appointment or for planned knee surgery

INTERVENTIONS:
Procedure: Exercise — Directional specific exercise
  Other Names: Repeated end range exercise
  Arms: Specific directional exercise
Procedure: Evidence based exercise — Quadriceps exercises and advice on aerobic exercises. Exercises are based on current evidence for the best exercises for osteoarthritic knee
  Other Names: step downs, resisted quadriceps, cycling, gym exercises
  Arms: Evidence based exercise

SUMMARY:
The purpose of the study is to explore if a subgroup of people with osteoarthritic knees can be identified using the McKenzie System of Mechanical Diagnosis and Therapy.

In the spine this subgroup, termed derangement,has been shown to respond rapidly to specific directional exercises.

The trial will explore whether these derangements in the knee respond to specific exercises compared to a control group with no exercises and non-derangement knees given general exercises.

DETAILED DESCRIPTION:
The Mechanical Diagnosis and Therapy (MDT) approach has been extensively used to classify and treat patients with spinal pain. Studies have shown this approach to be valid, reliable and able to predict outcome. Although the approach has been used for extremity joints there is no research on using this approach to classify individuals presenting with knee osteoarthritis.

An assessment tool that could potentially identify a subgroup of patients who would experience dramatic and rapid improvement to conservative care would be valuable.

Patients with an "osteoarthritic knee" diagnosis will be recruited after a consultation with an orthopaedic surgeon. Patients who consent to participate will be randomized into an intervention group and a control group. Baseline self reported function and pain will be collected. The control group will continue as planned on the waiting list for either a follow up orthopaedic consultation or for knee surgery. The intervention group will be assessed by one of three McKenzie credentialed therapist over 3 assessment sessions. The therapist will classify the patients as either having a "derangement" or not. Those classified as a derangement will have 2-3 follow up sessions and will be given direction specific exercises consistent with the principles of the McKenzie System over 2 weeks. Those patients who were not classified as derangements will be given 2-3 sessions of evidenced based osteoarthritis treatment consisting of strengthening exercises and advice on aerobic fitness exercise. At 2 weeks both groups will have baseline measures reassessed and will be discharged. Follow-up by telephone at 3 months and 1 year will reassess functional and pain measures.

Due to the high prevalence of knee osteoarthritis and the associated economic burden on our health care system it is important to investigate if physiotherapists are able to predict who will respond to conservative therapy. Classifying individuals with knee osteoarthritis into rapid responders or non responders to short-term physiotherapy treatment will allow more expensive medical evaluation and intervention to be directed to appropriate patients and avoid unnecessary treatment for patients likely to recover from less costly therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis
* Pain for longer than four months
* Knee X-ray/CT/MRI showing osteoarthritic changes
* Able to attend physiotherapy 2-3 times per week for 2 weeks
* Able to participate in exercise based therapy

Exclusion Criteria:

* Unable to provide informed consent
* Unable to understand written or spoken English
* Neurological conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Four item pain intensity measure (P4) | Change from Baseline in 3 months
  Measure of pain at different times of day as well as with activity on an eleven point scale from zero to ten

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 2 weeks, 3 months, 1 year
  Functional outcome measure specific for knee osteoarthritis with subscales of pain, symptoms, sport, function and quality of life
Intermittent and Constant Osteoarthritis Pain: Knee version (ICOAP) | Baseline, 2 weeks, 3 months, 1 year
  Measures nature of pain i.e. constant versus intermittent on a 5 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Rosedale, BSc, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Rosedale R, Rastogi R, May S, Chesworth BM, Filice F, Willis S, Howard J, Naudie D, Robbins SM. Efficacy of exercise intervention as determined by the McKenzie System of Mechanical Diagnosis and Therapy for knee osteoarthritis: a randomized controlled trial. J Orthop Sports Phys Ther. 2014 Mar;44(3):173-81, A1-6. doi: 10.2519/jospt.2014.4791. Epub 2014 Jan 22. PMID 24450370